CLINICAL TRIAL: NCT00671138
Title: A Phase 2a, Randomized, Double Blinded, Placebo Controlled, Study Evaluating Immunity and Gluten-sensitivity by Inoculating Celiac Disease Patients With the Human Hookworm Necator Americanus.
Brief Title: Inoculating Celiac Disease Patients With the Human Hookworm Necator Americanus: Evaluating Immunity and Gluten-sensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Princess Alexandra Hospital, Brisbane, Australia (Other)
Collaborators: The Broad Foundation (Other); Townsville Hospital (Other Government); James Cook University, Queensland, Australia (Other); Walter and Eliza Hall Institute of Medical Research (Other); Queensland Institute of Medical Research (Other)
Responsible Party: Principal Investigator, A James M Daveson, Doctor, Princess Alexandra Hospital, Brisbane, Australia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007/115; IBD-0214R
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Celiac Disease
Keywords: Celiac disease; Parasitic infections; necator americanus; Immunity
MeSH Terms: conditions — Celiac Disease; Parasitic Diseases | interventions — ASP-1 protein, Necator americanus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): Arm I will be inoculated with the human hookworm necator americanus at weeks 0 and 12.
  Interventions: Biological: Necator americanus
- II (Placebo Comparator): Arm II participants will receive and identical sham-inoculums comprising a diluted amount of 0.2ml McIlhenny & Co Tabasco Pepper Sauce®
  Interventions: Other: Sham inoculation

INTERVENTIONS:
Biological: Necator americanus — 10 necator americanus larvae will be inoculated at week 0 with a further 5 larvae inoculated at week 12
  Arms: I
Other: Sham inoculation — A diluted amount of McIlhenny & Co Tabasco Pepper Sauce will be applied via a gauze dressing at weeks 0 and 12.
  Arms: II

SUMMARY:
The disappearance of intestinal parasites from humans in developed countries may be responsible for the upsurge in many diseases including Celiac Disease, Crohn's, ulcerative colitis, asthma and hay fever. A parasite's survival relies on its ability to interfere with the host's immune response. The mechanisms employed to do this are similar to those required by a person to regulate against the so-called autoimmune disorders, diseases in which the system turns on itself. The investigators suspect that when parasites are excluded from the environment, some individuals become sufficiently self-reactive to develop an autoimmune disease. American researchers have successfully treated patients with Crohn's and ulcerative colitis using a pig whipworm (Trichuris suis). The investigators have undertaken a similar preliminary study using a human hookworm in Crohn's patients.

Using a small group of healthy people with celiac disease, the investigators will test if a human hookworm, Necator americanus, inhibits immune responsiveness to gluten. Celiac disease is a very common autoimmune-like disease (1% of Americans are affected although only a minority are aware they have the condition). In this condition, an individual becomes reactive to gluten, a protein in foods derived from wheat, barley, oats and rye.

What makes celiac disease such a good model for Crohn's disease is that similar immune changes are common to both, but in celiac disease the people are usually well, are not taking powerful immune suppressive drugs and the provocative antigens (the molecules that engage the immune system and provoke the disease) are known and can be excluded or introduced. As well as being of direct benefit to people with celiac disease, this study may give direction as to the potential of this parasite to manage inflammatory bowel disease.

People with proven celiac disease who live in Brisbane, a modern Australian city, will be invited to participate. Enrollment will require that the candidate has been avoiding gluten for six months.

The study is a blinded study (where the researchers and study subjects do not know who has gotten the parasites) aimed at comparing the disease activity and immunity after a controlled breach of the gluten-free diet in individuals with celiac disease, before and after hookworm infection. The disease severity and the immune system of celiac subjects before and after being inoculated with N. americanus will be examined using conventional and experimental investigations. This group's immunity will be compared to that of a group of matched, celiac control subjects (not infected with hookworm), before and after eating four pieces of standard white bread each day for three to five days. Twenty people, ten subjects per arm, will be recruited. Ten larvae initially, then five more after twelve weeks will be placed on the skin under a light dressing for thirty minutes.

The investigators aim to test whether the hookworm infection will change the immune processes and suppress gluten sensitivity in people with celiac disease. Outcomes to be measured will be those that reflect the activity of celiac disease.

DETAILED DESCRIPTION:
Background and aims: A number of lines of evidence suggest that the disappearance of helminths from human populations in developed countries may be responsible for the upsurge in autoimmune diseases, the so-called hygiene hypothesis. Using a small cohort of healthy subjects with quiescent celiac disease, our aim is to test if the ubiquitous hookworm (HW) of humans, Necator americanus, inhibits immune responsiveness to a gluten challenge (GC). As well as being of potential benefit to people with gluten intolerance, this study will provide the opportunity to undertake detailed investigation at the mucosal level of the host-parasite interaction, and the underlying immune response, and by extension, the potential of nematode infection to modulate the inflammatory response in IBD. Unlike experimental helminth infections in either animals genetically predisposed to colitis or in clinical IBD (where a range of complicating cofactors are present), this study addresses what happens in healthy humans who do not have a background of helminth exposure, and who are not currently compromised by either inflammation or immunosuppressive drugs.

Methods: Twenty healthy adults with well-documented celiac disease (DQ2 phenotype) compliant with a gluten-free (GF) diet for ≥ 6 months (based on history and a normal tissue transglutaminase [tTG]) will be recruited and randomly assigned to two groups of ten. Ten will be inoculated with hookworm (HW) larvae and 10 will serve as uninfected controls. Study subjects and Investigators will be blinded to allow comparison of disease activity and immune profiles. HW larvae will be cultured from feces supplied by a volunteer donor, previously infected for this purpose. Conventional endoscopy and biopsy will be performed twice per subject, before and after oral and rectal GCs (2x50g slices of wheat bread twice daily for 3-5 days and 6g of gluten in a 40ml slurry instilled into the rectum per endoscope, respectively). Rectal biopsy will be undertaken 4 hr and duodenal biopsy collected six days following GC; blood will be collected before and after acquiring hookworm infection and on day six following GC. Thus, four data sets will be accrued for comparison: ten GF celiac-subjects before HW infection; 10 GF celiac-s after HW infection; ten GC celiac-s before HW infection; and 10 GC celiac-s after HW infection.

Safety: A large body of observational data documenting the safety of experimental hookworm infection is available, both from our own and studies by others. Two of our researchers have maintained infections including occasional "top-up" inoculations for three years without ill effects.

Outcome Measures: These will include: subject symptom diary, full blood analysis, C-reactive protein, total and specific IgE and serum tryptase activity. The duodenal (Marsh classification) and rectal histology will be graded by a single pathologist. Goblet cells and mucosal T cells will be stained to aid quantification of responses. Peripheral blood mononuclear cells (PBMCs) and mucosal lymphocytes from intestinal biopsies will be grown ex vivo and challenged with gluten antigen immunodominant peptide (alpha-gliadin 57-73 Q65E, QLQPFPQPELPYPQPQS). Cell proliferation and cytokine profiles in response to HW and gluten antigens will be measured from PBMCs and intestinal biopsies. Varying the timing of the inoculations may provide worthwhile direction on the importance of the Th2 response only if there is a profound difference between newly established (Th2-dominant) versus mature (Th-neutral) parasite infections, as suggested by our earlier work with experimental human infections. Levels of transcription of genes of interest will be assessed using quantitative real time PCR and microarrays.

Outcomes: The null hypothesis is that Necator americanus does not change the immune process sufficiently to suppress gluten sensitivity in people with celiac disease. The measured outcomes reflect the activity of celiac disease, including the severity of mucosal inflammation, and the character and intensity of the immune processes. This study though is as much about IBD. Celiac disease is not IBD, but this model of IBD affords a previously unexplored opportunity to test quasi autoimmune responses in the duodenum and rectum to a specific antigen, one that can be introduced or excluded on demand. The immune profiling will focus on the characteristics that drive inflammation in IBD providing a clear insight as to the potential of helminths in Crohn's disease and ulcerative colitis.

Extension Study; Control patients invited to enroll in an extension of the study; each to be inoculated, challenged and investigated as per the original hookworm cohort (as above).

Low dose gluten challenge Study: This trial extension seeks to establish if hookworm infection might improve tolerance to small amounts of gluten in patients with celiac disease. The study is open. It utilises celiac patients already infected with hookworm and in whom the blood and mucosal baseline characteristics have been carefully documented. The gluten exposure will apply doses that have been demonstrated by others in a trial setting to be safe and well-tolerated. Effectiveness of hookworm infection to mitigate gluten intolerance will be measured by the quantifiable changes that occur in biopsies previously taken (pre-challenge) compared with tissue collected post-challenge.Histology will be performed as previously described. Biopsies are to be fixed in neutral buffered formalin, processed and carefully orientated and embedded in paraffin wax. Sections (3 μm) will be stained with haematoxylin and eosin (H&E) and immunostained with anti-CD8 (or anti-CD3 depending on availability) antibodies (Novocastra Laboratories Ltd). The intraepithelial lymphocytes (IELs) per 100 nucleated enterocytes (100NE) will be counted at 24 randomly selected sites between the villous tip and the base of the crypt (Vh/Cd) in each biopsy. Individual and collective outcomes on tissue collected after hookworm infection, but whilst on a gluten free diet, will be compared with those from tissue collected after the pasta challenge.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of celiac disease
* Positive tTG (IgA)or positive anti IgA gliadin or anti-endomysial antibody test.
* Marsh score ≥3 on small bowel biopsy (subtotal villous atrophy)
* Clinical, biochemical or histological improvement on gluten free diet.
* Compliance with a gluten-free diet for 6 months lead-in.
* Lifestyle & travel history indicative of a low risk for helminthic infection.
* Good general health not on immunomodifying agents.
* Ability to complete study
* Understand study & risks
* Social supports
* Workplace flexibility
* Normal tTG at enrollment (<10 dependent on serology)
* A HLA-DQ2 phenotype
* Negative fecal test for intestinal helminthes.
* Negative serological test for anti-strongyloides antibodies

Exclusion Criteria:

* Children (age < 18)
* Immunomodulating medication in 6 months pre-enrollment
* Oral or intramuscular/intravascular steroids
* Regular weekly use of aspirin
* Regular weekly use of NSAID
* Regular weekly use of COXII inhibitors
* Regular weekly use of statin medications
* Clinical history indicating a likely need to use an immune suppressive agent during the course of the study.
* Unmanaged risk of pregnancy
* Past history of infection with helminthes (other than a past history of infection with the pinworm, Enterobius vermicularis)
* History of insulin dependent diabetes mellitus or Addison's disease
* History of anaphylaxis or severe allergic reactions
* Having received a vaccine within the preceding 30 days
* Positive strongyloides serology
* Iron deficiency anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Duodenal histology (Marsh classification) and rectal histology | 21 weeks

SECONDARY OUTCOMES:
Peripheral blood mononuclear cells and mucosal lymphocytes will be grown ex vivo and challenged with gluten antigen immunodominant peptide. Cell proliferation and cytokine profiles will also be measured. | 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John T Croese, FRACP MD, Principal Investigator — The Townsville Hospital; A James M Daveson, MBBS, Study Director — Princess Alexandra Hospital; Alex Loukas, BSc Hon, PhD (UQ), Study Director — Queensland Institute of Medical Research; James McCarthy, MBBS FRACP PhD, Study Director — Queensland Institute of Medical Research; Robert Anderson, MB ChB BMedSc PhD FRACP, Study Director — Walter & Eliza Hall Institute of Immunology; Graeme Macdonald, MBBS FRACP PhD, Study Director — Princess Alexandra Hospital; Soraya Gaze, BSc PhD, Study Director — Queensland Institute of Medical Research; Rick Speares, MBBS PhD, Study Director — Anton Breinl Centre for Public Health and Tropical Medicine, James Cook University, Townsville; Andrew Clouston, MBBS (Qld) PhD (Qld) FRCPA, Study Director — Envoi Pathology; Andrew Pascoe, B. Pharm, B.Sc, MBBS, FRACP, Study Director — Princess Alexandra Hospital; Geoffrey Cobert, BSc PhD, Study Director — Queensland Institute of Medical Research; Dianne Jones, RN RM BAppSc, Study Director — Princess Alexandra Hospital; Sharon Cooke, RN, Study Director — The Townsville Hospital
Locations (3):
- Australia (3):
  - Queensland Institute of Medical Research, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Logan Hospital, Logan City, Queensland

REFERENCES:
- [Derived] Cantacessi C, Giacomin P, Croese J, Zakrzewski M, Sotillo J, McCann L, Nolan MJ, Mitreva M, Krause L, Loukas A. Impact of experimental hookworm infection on the human gut microbiota. J Infect Dis. 2014 Nov 1;210(9):1431-4. doi: 10.1093/infdis/jiu256. Epub 2014 May 3. PMID 24795483
- [Derived] Daveson AJ, Jones DM, Gaze S, McSorley H, Clouston A, Pascoe A, Cooke S, Speare R, Macdonald GA, Anderson R, McCarthy JS, Loukas A, Croese J. Effect of hookworm infection on wheat challenge in celiac disease--a randomised double-blinded placebo controlled trial. PLoS One. 2011 Mar 8;6(3):e17366. doi: 10.1371/journal.pone.0017366. PMID 21408161
- See also: Broad Medical Research Program Website — http://www.broadmedical.org